CLINICAL TRIAL: NCT03398265
Title: Treatment Navigation for Recently Released Prisoners With Opioid Use Disorder
Brief Title: Treatment Navigation for Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Caleb Banta-Green, Principal Research Scientist, Alcohol and Drug Abuse Institute, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000227
Record Dates: First submitted 2017-10-05; First posted 2018-01-12 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Initial discussion regarding opioid treatment options followed by 6 months of treatment navigation.
  Interventions: Behavioral: Treatment Navigation (Intervention)
- Control (Other): Referrals to treatment from corrections staff.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Treatment Navigation (Intervention) — Subjects in the intervention arm will begin a discussion with the interventionist about whether they are interested in treatment and medication choices for opioid use disorder. The interventionist will use a decision tool informed by the Substance Abuse and Mental Health Services Administration (SAMSHA) guide to medication assisted treatment in order to help make an informed decision about treatment choices. Once a decision is reached, the Treatment Navigator will communicate with the subject periodically to assist with entering treatment and help with locating other social services as needed within the community. The Treatment Navigator will emphasize getting into treatment as quickly as possible once a decision is made. The Treatment Navigator and the subject will continue communicating throughout the 6 month study period. Subjects will also receive overdose education and be offered take-home naloxone.
  Other Names: Treatment Navigation, Treatment Decision Making, Shared Decision Making
  Arms: Intervention
Other: Control — Subjects in the control arm will receive referrals from Department of Corrections (DOC) staff for treatment per DOC protocols. Subjects will not receive any treatment navigation or treatment decision making. Subjects will also receive overdose education and be offered take-home naloxone.
  Arms: Control

SUMMARY:
The investigators will conduct a pilot randomized controlled trial (RCT) study of 100 people with a history of opioid use disorder releasing to WA Department of Corrections (DOC) community corrections supervision in King County. Half of the subjects will receive treatment as usual (e.g. referral to treatment or outpatient drug counseling by DOC community corrections staff) and half will receive 6 months of intervention. The intervention involves treatment decision making, in which the study interventionists help subjects understand treatment choices, decide on the treatment that is best for them, get enrolled in treatment and remain in treatment. The study does not provide treatment, but works with treatment providers to facilitate access to care.

The aims of this study are to determine: 1) whether study procedures can be implemented with as designed, 2) whether offenders can be enrolled and maintained in the study, 3) which medications/treatment options subjects select and their experiences and satisfaction with the interventions, and 4) preliminary intervention effect size on outcomes of interest including recidivism, drug use, hospitalization, and treatment enrollment and retention.

ELIGIBILITY:
Inclusion Criteria:

1. Meets Diagnostic and Statistical Manual (DSM-5) criteria for opioid use disorder (at least 2 criteria) or were receiving treatment for opioid use disorder in the 12 months prior to incarceration.
2. Released to community corrections, not currently incarcerated.
3. Able to understand and provide informed consent.
4. Has access to phone (voice or text) or email to communicate with research staff.

Exclusion Criteria:

1. Under age 18 or over age 70 at time of recruitment.
2. Currently enrolled in an opioid treatment program using medications.
3. Has not used opioids (prescription type or heroin) in the past 6 months prior to incarceration.
4. Unwilling to allow access to medical or drug treatment records, criminal history or criminal activity records.
5. Inability to communicate in English verbally.
6. Inability to provide adequate contact information to assist with follow-up.
7. Not planning on being in King County or reporting to community corrections in King County for 6 months.
8. Violent or overtly hostile/threatening towards research staff.
9. Entering a controlled environment for 31 days or more in the next 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caleb Banta-Green, PhD, Principal Investigator — University of Washington
Locations (5):
- United States (5):
  - DOC Community Field Office, Auburn, Washington
  - DOC Community Field Office, Burien, Washington
  - DOC Community Field Office, Federal Way, Washington
  - DOC Community Field Office, Kent, Washington
  - DOC Community Field Office, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 125 people releasing from prison were identified by Washington Department of Corrections with notifications sent to local community corrections officers of their approximate release dates. Of the 125 people releasing from prison, 63 were approached for study participation. Of the 63 who were approached, 44 declined participation or were not opioid users. Of the remaining 19 who were assessed, 2 were ineligible and 17 were consented. Of the 17 who were consented, 15 were assigned to groups.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (7.3) | 37.1 (9.6) | 36.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15
Days of opioid use in last 30 days prior to incarceration [Mean (Standard Deviation); unit: days]
  Mean days used heroin | 24.8 (10.4) | 30 (0) | 27.8 (6.9)
  Mean days used prescription opioids | 19.8 (13.9) | 11.7 (15.9) | 16.8 (14.2)

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility
Description: The number of potentially eligible subjects self-referred or identified by Department of Corrections whom study staff were able to contact, screen, determine to be eligible and enroll in the study at Community Corrections facilities.
Time Frame: 6 months
Population: Of the 125 people releasing from prison, 63 were approached for study participation. Of the 63 who were approached, 44 declined participation or were not opioid users. Of the remaining 19 who were assessed, 2 were ineligible and 17 were consented. Of the 17 who were consented, 2 declined participation and15 were assigned to groups. The 15 assigned to groups were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 7 | 8
Participants | 7 | 8

2. Secondary Outcome: Criminal Activity
Description: The rate of arrests, charges and/or convictions for the comparison group versus the intervention group accounting for various potential residual confounders.
Time Frame: 1 month
Population: Criminal activity data were not obtainable and therefore analyses were not conducted.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Criminal Activity
Description: as for outcome 2
Time Frame: 6 months
Population: Criminal activity data were not obtainable and therefore analyses were not conducted.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hospitalizations
Description: The rate of hospitalizations for the comparison group versus the intervention group accounting for various potential residual confounders.
Time Frame: 1 month
Population: Hospitalization data were not obtainable and therefore analyses were not conducted.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Hospitalizations
Description: as for outcome 4
Time Frame: 6 months
Population: Hospitalization data were not obtainable and therefore analyses were not conducted.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Treatment Enrollment
Description: The rate of treatment enrollment for the comparison group versus the intervention group accounting for various potential residual confounders.
Time Frame: 1 month
Population: Treatment enrollment data were not obtainable and therefore analyses were not conducted.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Treatment Enrollment
Description: as for outcome 6
Time Frame: 6 months
Population: Because intervention feasibility was not demonstrated, treatment enrollment data were not obtained, and analyses were not conducted.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Relapse Prevention Medication Prescriptions
Description: The rate of medication initiation for the comparison group versus the intervention group accounting for various potential residual confounders.
Time Frame: 1 month
Population: Relapse prevention medication prescription data were not obtainable and therefore analyses were not conducted.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Relapse Prevention Medication Prescriptions
Description: as for outcome 8
Time Frame: 6 months
Population: Relapse prevention medication prescription data were not obtainable and therefore analyses were not conducted.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Nine months.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT03398265/Prot_SAP_001.pdf